CLINICAL TRIAL: NCT03298386
Title: Elderly Appropriate Treatment in Primary Care (EAT)
Acronym: TAPAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CIA : CNGE IRMG Association (Unknown); CNGE : Collège National des Généralistes Enseignants (Unknown); RMG : Institut de Recherche en Médecine Générale (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K170305; 2017- A01290 - 53 (Other: IDRCB)
Record Dates: First submitted 2017-07-31; First posted 2017-10-02 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Elderly; Polypharmacy
Keywords: Elderly; Multimorbidity; Polypharmacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group "STOPP/START" (Experimental): Training of General Practitioners with the tool STOPP/START Systematic medication review by GP with STOPP/START
  Interventions: Other: Systematic medication review with the STOPP/START tool
- Control group (No Intervention): Patient's usual care by the general practitioner (who will not be trained in the STOPP/START tool)

INTERVENTIONS:
Other: Systematic medication review with the STOPP/START tool — The STOPP / START tool includes a list of 42 substances / drug classes whose prescription could be discontinued based on specific criteria (81 STOPP criteria: Screening Tool of Older Person's Prescriptions) and a list of 34 clinical situations involving consideration of the usefulness of a new prescription (START criteria: Screening Tool to Action the Right Treatment).
  Arms: Intervention Group "STOPP/START"

SUMMARY:
The general practitioner (GP) is confronted, for a part of his clientele, with the management of patients suffering from multimorbidity, leading most often to a polypharmacy. It has five major consequences: increasing the number of inappropriate treatments, increasing the risk of potentially dangerous drug interactions, increasing the risk of contraindications associated with several concomitant pathologies, decreasing adherence to treatments by patients and the increased cost of care. Drug misuse in the elderly is particularly common, due to the age-related physiological changes and physiological alterations, with the consequent increase in the risk of adverse events, particularly hospitalizations. Several tools have been proposed to decrease morbimortality in elderly patients with polypharmacy. The studies concluded that the STOPP/START tool was the most structured, sensitive and had the most appropriate use format for clinical practice. However, there are currently no ambulatory studies demonstrating the impact of prescription revision with STOPP/START on the morbimortality of persons aged 75 years and over. This study aims to assess the effectiveness of an intervention targeting GPs to decrease morbimortality in elderly patients with polypharmacy. Volunteer GPs will be randomly assigned to either the intervention group or to usual care (control group) and they will be followed one year. The intervention consists in systematic medication review by GP with STOPP/START. In both groups, patient morbimortality will be measured at the end of the study.

DETAILED DESCRIPTION:
STOPP/START criteria for potential inappropriate prescribing in older people recognise the dual nature of inappropriate prescribing by including a list of potentially inappropriate medications (STOPP criteria) and potential prescribing omissions (START criteria).

ELIGIBILITY:
Inclusion Criteria:

* Patient 75 years of age or older
* With polypharmacy (≥ 5 medications)
* Not institutionalized
* Patient affiliated with the French health care system
* Oral consent given to participate in the study
* Patient who can be followed up 12 months
* Patient visiting the GP for any reason

Exclusion Criteria:

* Patient protected by law (under guardianship or curatorship)
* Having an estimated life expectancy of less than 12 months
* Participating in a therapeutic trial during the study period

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3032 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
A composite criterion: - percentage of unplanned hospitalization - percentage of death regardless of cause, - percentage of emergency department visit - percentage of institutionalization | at 12 months
  The primary outcome measure will be a composite criterion comprising unplanned hospitalization, death regardless of cause, emergency department visits and institutionalization after 12 months of follow-up.
  Unplanned hospitalization is defined as either hospitalization decided after a visit to the emergency department (whether the patient was sent by a doctor or not) or hospitalization decided on the same day by the general practitioner.

SECONDARY OUTCOMES:
Percentage of unplanned hospitalization | at 12 months
Percentage of death regardless of cause | at 12 months
Percentage of emergency department visits | at 12 months
Percentage of institutionalization | at 12 months
Percentage of loss of autonomy | at 12 months
  The loss of autonomy at 12 months defined by the loss of at least one activity of the daily living (ADL) between the intervention and 12 months of follow-up.
Decrease in the number of drugs on the prescription (%) | at 12 months
  The decrease in the number of drugs on the prescription (Polypharmacy decrease) between baseline and 12 months of follow-up
Percentage of falls | at 12 months
Percentage of recommendations followed | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julien Le Breton, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Clinical Epidemiology and Ageing (CEpiA) EA7376 Faculté de Médecine, Université Paris Est Créteil (UPEC), Créteil, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. Proposals should be directed to ASSISTANCE PUBLIQUE HOPITAUX DE PARIS [AP-HP], Department for Clinical Research, Innovation (DRCI) represented by Mr Milan LAZAREVIC,Director . To gain access, data requestors will will need to sign a data transfer agreement with the sponsor.

REFERENCES:
- [Background] O'Mahony D, O'Sullivan D, Byrne S, O'Connor MN, Ryan C, Gallagher P. STOPP/START criteria for potentially inappropriate prescribing in older people: version 2. Age Ageing. 2015 Mar;44(2):213-8. doi: 10.1093/ageing/afu145. Epub 2014 Oct 16. PMID 25324330
- [Background] Dalleur O, Spinewine A, Henrard S, Losseau C, Speybroeck N, Boland B. Inappropriate prescribing and related hospital admissions in frail older persons according to the STOPP and START criteria. Drugs Aging. 2012 Oct;29(10):829-37. doi: 10.1007/s40266-012-0016-1. PMID 23044639
- [Background] Gallagher PF, O'Connor MN, O'Mahony D. Prevention of potentially inappropriate prescribing for elderly patients: a randomized controlled trial using STOPP/START criteria. Clin Pharmacol Ther. 2011 Jun;89(6):845-54. doi: 10.1038/clpt.2011.44. Epub 2011 Apr 20. PMID 21508941
- [Background] Dalleur O, Boland B, Losseau C, Henrard S, Wouters D, Speybroeck N, Degryse JM, Spinewine A. Reduction of potentially inappropriate medications using the STOPP criteria in frail older inpatients: a randomised controlled study. Drugs Aging. 2014 Apr;31(4):291-8. doi: 10.1007/s40266-014-0157-5. PMID 24566877
- [Background] Frely A, Chazard E, Pansu A, Beuscart JB, Puisieux F. Impact of acute geriatric care in elderly patients according to the Screening Tool of Older Persons' Prescriptions/Screening Tool to Alert doctors to Right Treatment criteria in northern France. Geriatr Gerontol Int. 2016 Feb;16(2):272-8. doi: 10.1111/ggi.12474. Epub 2015 Mar 21. PMID 25809727
- [Derived] Guellich A, Oubaya N, Cogneau J, Lacoin F, Clerc P, Audureau E, Le Breton J. Identifying patterns of multimorbidity, polypharmacy and frailty in the elderly: a clustering analysis of baseline data from a French, randomised, controlled trial in primary care. BMJ Open. 2025 Jun 27;15(6):e083584. doi: 10.1136/bmjopen-2023-083584. PMID 40578876